CLINICAL TRIAL: NCT06718725
Title: An Artificial Intelligence System for Rapid Onsite Cytologic Pathology Evaluation（ROSE） of Endoscopic Ultrasound-guided Fine-needle Aspiration (EUS-FNA) Sample: a Prospective, Multicenter, Diagnostic Study.
Brief Title: An Artificial Intelligence System for ROSE of EUS-FNA Sample: a Prospective, Multicenter, Diagnostic Study.
Acronym: ROSE，EUS-FNA
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Taian City Central Hospital (Other); Qilu Hospital of Shandong University (Qingdao) (Other); Shandong Provincial Hospital (Other Government); Liaocheng People's Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Binzhou People's Hospital (Other); Binzhou Medical University (Other); 960th Hospital of PLA (Unknown); Yidu Central Hospital of Weifang (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024SDU-QILU-1
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-09

CONDITIONS: The Malignant Lesions and Non-malignant Lesions of Pancreas, Bile Duct, Liver and Lymph Node

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — cytopathological slide images from patients who underwent EUS-FNA and ROSE
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing EUS-FNA and ROSE: Patients ≥18 years with pancreatic, bile duct, hepatic, or lymph node lesions accepted EUS-FNA and ROSE.
  Interventions: Diagnostic Test: ROSE-AI system

INTERVENTIONS:
Diagnostic Test: ROSE-AI system — The cytopathological slide images of the patients' ROSE samples will be identified by the ROSE-AI system.

SUMMARY:
This is an observational study with a prospective, multicenter, disgnostic design. An artificial intelligence system named ROSE-AI system was developed using cytopathological slide images taken by microscope camera or smartphone of pancreas, bile duct, liver and lymph node, collected retrospectively from patients who underwent EUS-FNA and ROSE, and the performance of ROSE-AI system was validated in the datasets collected prospectively.This study aims to assist endoscopists in conducting rapid on-site cytopathology evaluations during EUS-FNA without the presence of cytopathologists. In addition, the diagnostic field was compared between the cytopathologists and ROSE-AI system, endoscopists with or without ROSE-AI system.

ELIGIBILITY:
Inclusion Criteria:

1. the patient age ≥18 years accepted EUS-FNA+ROSE.
2. agree to participate in the research and be able to sign written informed consent.

Exclusion Criteria:

1. uncorrectable coagulopathy (PTT >50 seconds or INR >1.5) and/or uncorrectable thrombocytopenia (platelet count <50 × 109 /L).
2. patients who were too clinically ill to undergo an EUS examination.
3. lesions that were deemed inaccessible for EUS-guided sampling.
4. unsuccessful EUS-FNA (e.g., failure to obtain an adequate specimen, patient intolerance, intraoperative accidents, etc.).
5. Patients with unqualified ROSE smear.
6. Patients who underwent biopsy during EUS-FNA but did not receive a definitive pathological diagnosis or pathological report.
7. pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with pancreatic, bile duct, hepatic, or lymph node lesions undergoing EUS-FNA and ROSE from the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
the accuracy, sensitivity and specificity of the ROSE-AI system in identifying malignant/non-malignant ROSE samples | During procedure
  The primary outcome of the study is to evaluate the performance of the ROSE-AI system in identifying the malignant/non-malignant ROSE samples of pancreatic, bile duct, hepatic and lymph node based on both images taken by microscope camera and smartphone, and comparing the performance between the ROSE-AI system and endoscopists, cytopathologists.

SECONDARY OUTCOMES:
comparing the diagnostic performance between endoscopists with ROSE-AI system and without ROSE-AI system | During procedure
  A cross-over human-AI contest using images of the prospective testing dataset will be performed. The diagnostic performance of endoscopists with ROSE-AI system and without ROSE-AI system will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No